CLINICAL TRIAL: NCT04399304
Title: Safety of Bilateral HTO: One-Stage vs.Two-Stage: A Randomized Controlled Study
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Orkhan Aliyev, MD, Resident Doctor in Orthopaedic Surgery, Bezmialem Vakif University
Other Study IDs: 45446446-020-5169
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Gonarthrosis; Primary; Varus Gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Simultaneous: One-stage bilateral high tibial osteotomy
  Interventions: Procedure: simultaneous bilateral high tibial osteotomy
- Staged: Two-stage bilateral high tibial osteotomy
  Interventions: Procedure: Staged bilateral high tibial osteotomy

INTERVENTIONS:
Procedure: simultaneous bilateral high tibial osteotomy — One-stage simultaneous bilateral high tibial osteotomy
  Groups: Simultaneous
Procedure: Staged bilateral high tibial osteotomy — Two-stage bilateral high tibial osteotomy
  Groups: Staged

SUMMARY:
In this study, bilateral simultaneous high tibial osteotomy (HTO) was compared with staged bilateral HTO in terms of complications. We did not use any grafts to support the osteotomy line and the patients were mobilized immediately with a full load on a postoperative day 1. And our hypothesis is that bilateral simultaneous applications are safe in comparison to the staged ones in terms of complications.

DETAILED DESCRIPTION:
Knee osteoarthritis is the most common orthopedic chronic disease, and varus knee abnormalities can often be related. The load from the medial tibiofemoral joint increases significantly in varus alignment disorder and it plays an important role in the structural progression of knee osteoarthritis. Varus malalignment and patients with medial tibiofemoral disease comprise a common patient subset. The probability of progressing to severe disease is 3 to 4 times higher in these patients compared to those with a neutral knee alignment. Although the long-term results of high tibial osteotomy are well documented, but data on bilateral simultaneous HTO are insufficient. In general, staged surgery is preferred in bilateral cases due to the difficult rehabilitation, healing of the osteotomy line, and complications related to surgery. Advances in post-surgical rehabilitation have been made due to increased confidence in stability due to improvements in the technology of plates.The advantages of an bilateral simulatneous HTO is single administration of anesthesia, total shortening of the hospitalization periof and reduced costs.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral primary genu varus gonarthrosis

Exclusion Criteria:

* Secondary gonarthrosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bilateral genu varus gonarthrosis operated by the tertiary step hospital high-volume knee surgeons
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Complications | 2 year
  Total complications rate

SECONDARY OUTCOMES:
Radiologic assesment | 2 year
  Changes in corrections degree

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No